CLINICAL TRIAL: NCT03114813
Title: Beta-blocker Stratification Using Quantitative MRI Techniques to Assess Portal Pressure and Response to Treatment in Patients With Portal Hypertension
Brief Title: Can MRI Evaluate Beta-blocker Response in Portal Hypertension?
Acronym: B-SMaRT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Nottingham (Other)
Collaborators: University Hospitals of Derby and Burton NHS Foundation Trust (Other); Nottingham University Hospitals NHS Trust (Other); University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 16049
Record Dates: First submitted 2017-01-13; First posted 2017-04-14 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-04

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Varix, Esophageal
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal; Esophageal and Gastric Varices | interventions — Carvedilol; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Clinically indicated primary prophylaxis: Approach all those who have had a portal pressure measurement (HVPG) as part of their routine clinical care.
  At baseline participants will consent to have an additional MRI scan before undergoing clinical screening Endoscopy.
  All participants found to have oesophgeal varices that require primary prophylaxis, will be started on Carvedilol 6.25mg.
  After 1 week, participants will return for dose optimisation
  After 4-12 weeks of treatment, participants will have:
  * repeat one hour MRI scan
  * repeat HVPG to evaluate treatment response
  Interventions: Drug: Carvedilol; Other: MRI scan; Procedure: Hepatic Venous Pressure Gradient (HVPG)

INTERVENTIONS:
Drug: Carvedilol — Non-selective beta-blocker as per routine clinical care
Other: MRI scan — One hour non-invasive MRI scan
Procedure: Hepatic Venous Pressure Gradient (HVPG) — Second HVPG to evaluate treatment response

SUMMARY:
Aim:

To test if MRI can detect meaningful changes in portal pressure in the liver to assess whether treatment with beta-blockers has worked.

Liver Disease:

Most people with liver disease do not have symptoms. Over time they develop 'cirrhosis' - severe liver scarring. In the United Kingdom deaths due to cirrhosis have doubled over the last decade, because of increasing rates of alcohol consumption and obesity, while heart, kidney, lung diseases, strokes and cancer fatalities have fallen.

Portal pressure:

Cirrhosis causes increased pressure within the liver and changes in the circulation leading to the development of varicose veins in the gullet and stomach called 'varices'. Varices bleed easily, leading to emergency situations that can be life threatening. However, if the increased pressure within the liver (portal pressure) is detected early, then treatment can prevent variceal bleeding. The only test we have to predict prognosis and treatment success in someone with cirrhosis is by measuring the portal pressure.

Measuring portal pressure:

Currently the only existing test to measure portal pressure is to pass a pressure sensor through a vein in the neck, down into the liver. This is called the hepatic venous pressure gradient (HVPG) measurement. The HVPG measurement is disliked by patients because it is an invasive procedure. It is also expensive and not widely available. Hence, patients with cirrhosis need to have regular camera tests (endoscopies) to look for varices.

How can you treat varices?

Two options;

1. With tablets to lower the pressure (beta-blockers)
2. Endoscopy treatment (banding)

Both have advantages and disadvantages;

* Beta-blockers only lower the portal pressure in about half of those that take them, with some evidence they may also have a protective effect against infections from the bowel by increasing the speed of bowel motion
* Treating the varices with endoscopy requires several endoscopies and can lead to life-threatening bleeding.

Most patients are therefore given beta-blockers and monitored closely to see if they work.

Why does it matter?

Beta-blockers can cause side effects (e.g. fainting) that are unpleasant enough to make up to one third of patients stop taking them. Beta-blockers only reduce the portal pressure in half of patients. The remaining patients are exposed to potential side effects and possible harm in those with the most advanced liver disease. These patients may still have a life-threatening bleed as the varices have not been adequately treated. There is a desperate need to discover whether the portal pressure changes with treatment (such as with beta-blockers) without invasive tests across the NHS.

Proposed study:

Researchers in Nottingham have shown MRI can be used as an accurate marker of portal pressure with just one scan. To be useful to patients, doctors and researchers, this study will investigate whether MRI can detect meaningful changes in portal pressure after treatment with beta-blockers. This study has been designed with patient and public involvement (PPI) integrated throughout. A focus group shaped the study design and committed to collaborate in developing patient materials, recruitment, retention and dissemination.

All patients who have HVPG will be given information about the study.

Study Visit 1

* One hour MRI scan
* Endoscopy to identify varices

  * If varices are present the patient will be started on beta-blockers and invited to visit 2
  * If there are no varices, patients will return to regular follow up with the liver team

Study Visit 2 (after one week)

* Assess side effects, blood pressure and pulse
* Increase dose of beta-blocker as appropriate

Study Visit 3 (after 4-12 weeks)

* One hour MRI scan
* Repeat HVPG measurement

Treatment success is determined by the second HVPG measurement. If beta-blockers are working they will be continued. If not, the patient will have treatment with endoscopy. This represents the ideal pathway which is more personalised than current standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patients of more than 18 and less than 85 years of age
* Patients who have had HVPG measurements within the last 12 weeks.
* Underlying portal hypertension due to chronic liver disease - alcoholic liver disease, non-alcoholic fatty liver disease (NAFLD), chronic hepatitis B or C and haemochromatosis.
* Patients investigated with a clinical suspicion of portal hypertension, but have normal portal pressures on HVPG measurements.
* Ability to consent to participate in the study.
* Patients already on NSBBs who have stopped treatment for two weeks

Exclusion Criteria:

* Unable to give informed consent
* Patients with underlying diseases which are NOT related to alcohol excess, NAFLD, chronic hepatitis B, C or haemochromatosis.
* Pregnant women.
* Absolute contraindications for MRI (including participants with metal in/around the eyes)
* Absolute contraindications for NSBBs (allergy, presence of asthma)
* Patients currently on NSBBs or nitrates (can be included if withheld for two weeks)
* mean arterial pressure <55 mm Hg or pulse < 50 beats per minute at baseline

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with HPVG
Sampling Method: Non-Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-07 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Kappa agreement between quantitative MRI estimates of HVPG (modelled by liver T1 and splenic artery velocity) and HVPG to stratify treatment response to beta-blockers in patients requiring primary prophylaxis for oesophageal varices. | Within 12 weeks of starting treatment with beta-blockers

SECONDARY OUTCOMES:
Validate univariate and multivariate quantitative MRI measures (structural, haemodynamic) associated with portal pressure at a field strength of 3 Tesla (in particular previously published model with T1 and splenic artery velocity) | At study visit 1
Characterise the correlation between MR elastography measures of liver stiffness at 3 Tesla with T1 relaxation time based structural changes | At study visit 1

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - NIHR Nottingham Biomedical Research Centre, Nottingham, Nottinghamshire
  - University of Nottingham, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: NIHR Nottingham Digestive Diseases Biomedical Research Unit website — https://nddcbru.org.uk